CLINICAL TRIAL: NCT01615497
Title: Computer Based Training in Cognitive Behavioral Therapy Web-based Delivery of CBT4CBT for Alcohol
Brief Title: Web-based CBT4CBT for Alcohol
Acronym: CBT4CBT Etoh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1204010157; R21AA021405-01 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Abuse or Dependence
Keywords: cognitive behavior therapy; computer assisted instruction; alcohol abuse therapy; educational resource design and development
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Treatment as Usual (TAU) (Active Comparator): Treatment that would normally be received at the clinic typically consisting of individual or group counseling sessions focusing on alcohol and substance abuse.
  Interventions: Behavioral: Standard Treatment as Usual (TAU)
- Web-based CBT4CBT for alcohol plus TAU (Experimental): A computerized program that teaches skills for stopping drug and alcohol use by increasing coping skills such as how to understand patterns of drug use, coping with cravings, etc. plus standard treatment as usual.
  Interventions: Behavioral: Web-based CBT4CBT for alcohol plus TAU
- Web-based CBT with minimal clinical contact (Active Comparator): A computerized program that teaches skills for stopping drug and alcohol use by increasing coping skills such as how to understand patterns of drug and alcohol use, coping with cravings, etc. plus 10 minute check in with clinician.
  Interventions: Behavioral: Web-based CBT with minimal clinical contact

INTERVENTIONS:
Behavioral: Standard Treatment as Usual (TAU) — Treatment normally offered at this clinic which could include individual or group alcohol and drug counseling sessions one time per week lasting one hour each time.
  Arms: Standard Treatment as Usual (TAU)
Behavioral: Web-based CBT4CBT for alcohol plus TAU — Subjects work with a computerized program that teaches skills for stopping alcohol and drug use and increasing coping skills. Computerized sessions are one time per week and last about one hour per session. Plus TAU
  Arms: Web-based CBT4CBT for alcohol plus TAU
Behavioral: Web-based CBT with minimal clinical contact — Subjects work with a computerized program that teaches skills for stopping alcohol and drug use and increasing coping skills. Computerized sessions are one time per week and last about one hour per session. Plus 10 minute check in with clinician.
  Arms: Web-based CBT with minimal clinical contact

SUMMARY:
The investigators are conducting a randomized clinical trial of our new web-based version of the CBT4CBT (Computer Based Training for Cognitive Behavioral Therapy) program specifically designed for alcohol to evaluate its effectiveness relative to standard outpatient counseling at the Substance Abuse Treatment Unit (SATU). The computer-based training program (CBT4CBT) focuses on teaching basic coping skills, presenting examples of effective use of coping skills in a number of realistic situations in video form, and providing opportunities for patients to practice and review new skills while receiving substance abuse treatment.

DETAILED DESCRIPTION:
Ninety alcohol using individuals seeking treatment at the Substance Abuse Treatment Unit (SATU) of the Connecticut Mental Health Center will be randomized to (1) standard outpatient counseling at SATU (typically consisting of weekly group counseling), (2) standard outpatient counseling plus web-based CBT, or (3) web-based CBT4CBT with minimal clinical monitoring. Treatments will be delivered over an 8-week period with a six-month follow-up after termination of the study treatments. The primary outcome measures will be reduction in alcohol use (frequency of alcohol use by time, confirmed by urine toxicology screens and breathalyzers). Secondary outcomes will include treatment utilization and cost, several measures intended to detect whether web-based CBT4CBT retains key characteristics of traditional clinician-administered CBT (e.g., acquisition of coping skills, use of change strategies), participant characteristics which will be evaluated as potential moderators of outcome, as well as participant satisfaction and treatment credibility.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older.
* Are applying for outpatient, non-agonist substance abuse treatment at SATU.
* Meet current DSM-IV criteria for alcohol abuse or dependence.
* Are sufficiently stable for 8 weeks of outpatient treatment.
* Can commit to 8 weeks of treatment and are willing to be randomized to treatment
* Are willing to provide locator information for follow-up.
* Are fluent in English and have a 6th grader or higher reading level

Exclusion Criteria:

* Have an untreated bipolar or schizophrenic disorder.
* Who have a current legal case pending such that incarceration during 8-week protocol is likely.
* Are physically dependent on alcohol, opioids or benzodiazepines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction in alcohol use | 8 weeks

SECONDARY OUTCOMES:
Subjects ability to demonstrate coping skills through a computerized role-playing evaluation and homework | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- Substance Abuse Treatment Unit (SATU), New Haven, Connecticut, United States

REFERENCES:
- [Derived] Kiluk BD, Devore KA, Buck MB, Nich C, Frankforter TL, LaPaglia DM, Yates BT, Gordon MA, Carroll KM. Randomized Trial of Computerized Cognitive Behavioral Therapy for Alcohol Use Disorders: Efficacy as a Virtual Stand-Alone and Treatment Add-On Compared with Standard Outpatient Treatment. Alcohol Clin Exp Res. 2016 Sep;40(9):1991-2000. doi: 10.1111/acer.13162. Epub 2016 Aug 4. PMID 27488212